CLINICAL TRIAL: NCT00423358
Title: Treatment of Hypovitaminosis D in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-0011; K23AR050995 (NIH)
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-07

CONDITIONS: Rheumatoid Arthritis; Hypovitaminosis D
Keywords: rheumatoid arthritis; hypovitaminosis D; bone turnover; ergocalciferol
MeSH Terms: conditions — Arthritis, Rheumatoid; Vitamin D Deficiency | interventions — Vitamin D; Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D (Active Comparator): ergocalciferol 50,000 IU Twice monthly
  Interventions: Dietary Supplement: Vitamin D
- placebo (Placebo Comparator): matching placebo tablet
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Ergocalciferol 50,000 IU loading dose then twice monthly for one year
  Other Names: ergocalciferol
  Arms: vitamin D
Dietary Supplement: placebo — matching placebo
  Arms: placebo

SUMMARY:
This study recruits individuals with rheumatoid arthritis (RA) and low vitamin D concentrations. Subjects are dosed with vitamin D or placebo for one year. Primary outcome is change in bone turnover markers, additionally, bone mineral density and parameters of RA status are evaluated throughout the study.

DETAILED DESCRIPTION:
Osteoporosis is twice as common in people with rheumatoid arthritis (RA), compared to age and gender-matched controls [1, 2]. Hypovitaminosis D can contribute to osteoporosis pathogenesis by decreasing calcium absorption, leading to a decline in serum ionized calcium, a rise in parathyroid hormone levels and upregulation of osteoclast activity, leading to loss of calcium from the skeleton. Hypovitaminosis D is also common in patients with rheumatoid arthritis [3-5], making it an appealing target to potentially improve health in both RA and osteoporosis.

Vitamin D has theoretic potential to modulate RA disease activity, based on the presence of vitamin D receptors in lymphocytes, macrophages, chondrocytes, and synovial cells [6]. Vitamin D, given as the bioactive metabolite 1,25(OH)2D, ameliorates disease activity in murine models of RA [7, 8]. However, few studies have evaluated the effect of vitamin D on RA disease activity in humans. Two three month open-label studies reported that vitamin D reduced RA disease activity [9] and pain levels [10]. By contrast, an eight-week open-label study [11] reported no reduction in swollen joint counts, inflammatory markers or cytokine levels after vitamin D therapy. The only double-blind, placebo-controlled trial published thus far [12] found no significant effect of vitamin D on RA disease activity, but was limited by the lack of hypovitaminosis D as a criterion for study entry. Indeed, at baseline subjects' mean 25(OH)D levels indicated vitamin D repletion, potentially explaining the null effect of vitamin D on RA disease activity.

Three studies have evaluated the effect of vitamin D on bone mineral density (BMD) in patients with RA [13-15]. Researchers [14] randomized 96 subjects with RA to vitamin D (500 IU/day) and calcium (1000 mg/day) or placebo for two years; vitamin D and calcium therapy modestly increased BMD in the spine and hip. In another study [15], 20 subjects randomized to daily calcium and 1 α-hydroxyvitamin D for up to 24 months experienced similar declines in radius and spine BMD compared to 15 controls [15]. Likewise, vitamin D and calcium did not prevent bone loss in a prospective cohort study of patients with RA [13]. However, none of the studies required hypovitaminosis D as an entry criterion, vitamin D repletion to 25(OH)D levels > 32 ng/ml were not evaluated [13, 14] or achieved [15], and low doses of vitamin D were administered, potentially limiting skeletal benefits of this therapy.

We hypothesized that correction of hypovitaminosis D in subjects with RA would decrease parathyroid hormone (PTH), increase BMD, improve functional capacity and down-regulate inflammatory cytokine production, thereby diminishing disease activity. Vitamin D is inexpensive and widely available. If proven beneficial, vitamin D might become a mainstay of therapy for subjects with RA.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatology

Exclusion Criteria:

* Bisphosphonate therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-02; Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Hansen, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Hansen KE, Jones AN, Lindstrom MJ, Davis LA, Engelke JA, Shafer MM. Vitamin D insufficiency: disease or no disease? J Bone Miner Res. 2008 Jul;23(7):1052-60. doi: 10.1359/jbmr.080230. PMID 18302509
- [Result] Hansen KE, Bartels CM, Gangnon RE, Jones AN, Gogineni J. An evaluation of high-dose vitamin D for rheumatoid arthritis. J Clin Rheumatol. 2014 Mar;20(2):112-4. doi: 10.1097/RHU.0000000000000072. No abstract available. PMID 24561419

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 9 | 15
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12) | 53 (11) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Parathyroid Hormone Level
Description: Serum parathyroid hormone level
Time Frame: 1 Year
Population: Subject data were analyzed using the intent to treat approach.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Vitamin D, n=11: ergocalciferol 50,000 IU Twice monthly
  Vitamin D: Ergocalciferol 50,000 IU loading dose then twice monthly for one year
- Placebo, n=11: matching placebo tablet
  placebo: matching placebo
Arm/Group | Vitamin D, n=11 | Placebo, n=11
Number analyzed (Participants) | 11 | 11
pg/mL | 19 (11) | 20 (11)

2. Secondary Outcome: Bone Mineral Density
Description: one year change in mean total hip BMD
Time Frame: 1 Year
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Vitamin D, n=11 | Placebo, n=11
Number analyzed (Participants) | 11 | 11
g/cm2 | 0.970 (0.140) | 1.151 (0.168)

3. Secondary Outcome: Short Form 36 Survey
Description: 12 month score for physical function domain of SF36 survey; scale 0 to 100 with 0 indicating worst disability and 100 indicating best physical function
Time Frame: 1 Year
Population: Intent to treat analysis
Measure: Mean (95% Confidence Interval); unit: units from 0 (worst) to 100 (best)
Arm/Group | Vitamin D, n=11 | Placebo, n=11
Number analyzed (Participants) | 11 | 11
units from 0 (worst) to 100 (best) | 39.1 [34.0 to 44.4] | 47.7 [42.5 to 52.9]

ADVERSE EVENTS:
Time Frame: Adverse events were queried through specific and open ended questions at each study visit. All AEs after randomization were counted and reported.
Arm/Group | Vitamin D, n=11 | Placebo, n=11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D, n=11 (N=11) | Placebo, n=11 (N=11)
GI (Gastrointestinal disorders) | 1 (1) | 0 (0) — One participant in the treatment arm reported stomach cramping and constipation that resolved within two weeks of stopping calcium supplements, despite continuation of vitamin D therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No